CLINICAL TRIAL: NCT05813353
Title: Usability Study of the BAMCOG Followed by Concurrent Validation of the BAMCOG With the MoCA as a Monitoring Instrument for Perioperative Cognitive Function
Brief Title: Pre- and Post TAVI Cognitive Functioning and Intraoperative Carotid Flow Measurements
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Mariska te Pas, Drs. Mariska te Pas, Catharina Ziekenhuis Eindhoven
Other Study IDs: nWMO-2020.106
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Impairment; Older People--Abuse of; Aortic Stenosis, Severe
MeSH Terms: conditions — Cognitive Dysfunction; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose:

1. Measuring and optimize the usability of the BAMCOG (games to measure cognitive functioning)
2. Concurrent validation of BAMCOG with MoCA to see if BAMCOG can serve as a monitoring instrument/screener
3. Determination of carotid flow/cerebral blood flow pre- and post implant of prosthesis of aortic valve by ultrasound doppler measurements

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old
* Scheduled for TAVI surgery
* Able to play games on a tablet
* For usability part > MoCA score of 26 or higher
* Near native dutch speaker

Exclusion Criteria:

* Mental disorder (unable to play games)
* Alcohol abuse (women <15 and men >22 alcoholic drinks/week)
* No informed consent
* Atrial fibrillitation (for ultrasound doppler)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing TAVI surgery
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Usability of BAMCOG | 3 months preoperative
Concurrent validation of BAMCOG with MoCA | 3 months preoperative - 3 months postoperative
Cerebral perfusion/carotid flow measurements | Peroperative

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, Netherlands